CLINICAL TRIAL: NCT06644391
Title: Enhancing Diagnostic Accuracy in Fracture Identification on Musculoskeletal Radiographs Using Deep Learning
Status: Completed | Type: Observational
Sponsor: Carebot s.r.o. (Industry)
Responsible Party: Sponsor
Other Study IDs: CB-BONES-01-FM
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Fractures; Musculoskeletal
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiographs Analyzed Using AI and Radiologist Review: This cohort consists of 600 radiographs collected from pediatric and adult patients, aged 1 to 99 years, who underwent X-ray imaging for musculoskeletal conditions. The radiographs include various body parts such as the foot, ankle, knee, hand, wrist, elbow, shoulder, and pelvis. Fractures were present in 95 cases, while 453 cases showed no fractures.
  Interventions: Diagnostic Test: Carebot AI Bones

INTERVENTIONS:
Diagnostic Test: Carebot AI Bones — The use of a deep learning-based artificial intelligence software, Carebot AI Bones version 1.2.2, designed to aid in the detection of fractures on musculoskeletal radiographs. The AI model analyzes digital X-ray images to identify fractures, highlighting areas of interest with bounding boxes.

SUMMARY:
This retrospective study aims to evaluate the effectiveness of artificial intelligence (AI) in identifying fractures on musculoskeletal X-rays. By comparing the performance of a deep learning AI model with that of experienced radiologists, we seek to understand how AI can help improve fracture detection accuracy in clinical settings. The study analyzed 600 X-rays from both pediatric and adult patients, focusing on identifying fractures across different body parts, including the foot, ankle, knee, hand, wrist, and more. The findings show that integrating AI can increase radiologists' sensitivity in detecting fractures, potentially improving patient outcomes by reducing the number of missed injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1 year or older.
* Musculoskeletal X-rays available in Digital Imaging and Communications in Medicine (DICOM) format.
* At least one digital plain radiograph of an appendicular body part, including the foot, ankle, knee, hand, wrist, elbow, shoulder, or pelvis.

Exclusion Criteria:

* Poor radiographic quality that precludes human interpretation.
* Radiographs of the lumbar, thoracic, and cervical spine, or facial/nasal bones.
* Radiographs that do not meet the inclusion criteria for appendicular body parts.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study includes a retrospective cohort of pediatric and adult patients who underwent musculoskeletal radiographs between March 20 and May 8, 2023, in a single-center hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity of AI Model Compared to Radiologists in Fracture Detection on Musculoskeletal X-rays | From March 2023 to May 2023 (Retrospective analysis period)
  This outcome measures the sensitivity of the AI model (Carebot AI Bones 1.2.2) in detecting fractures on musculoskeletal X-rays, compared to the sensitivity of radiologists with varying levels of experience. Sensitivity is calculated as the proportion of true positive fracture cases identified by the AI model and radiologists out of all confirmed fracture cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Nemocnice ve Frýdku-Místku, p.o., Frýdek-Místek, Moravskoslezský kraj, Czechia

IPD SHARING:
Plan to Share IPD: No
Due to privacy concerns and the retrospective nature of the study, individual participant data (IPD) will not be shared. Data collected contains sensitive medical information that is protected under confidentiality agreements and GDPR regulations.